CLINICAL TRIAL: NCT07283562
Title: Efficacy and Safety of Gastrodin Acupoint Injection as an Adjunctive Therapy for Sensorineural Hearing Loss With Vertigo: A Randomized Controlled Trial
Brief Title: Gastrodin Acupoint Injection for Sensorineural Hearing Loss With Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Wu Yuan, Doctor, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022072
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Sensorineural Hearing Loss; Vertigo
MeSH Terms: conditions — Hearing Loss, Sensorineural; Vertigo | interventions — gastrodin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAI Group (Experimental): Participants received conventional therapy plus Gastrodin Acupoint Injection (GAI).
  Interventions: Drug: Gastrodin Injection
- Control Group (Active Comparator): Participants received conventional therapy only.
  Interventions: Drug: Conventional Therapy

INTERVENTIONS:
Drug: Gastrodin Injection — 0.5 mL (25 mg) gastrodin injected into selected acupoints alternating between Set A (Tinggong, Tinghui, Yifeng) and Set B (Baihui, Taichong, Neiguan, Shenmen) once every two days for 4 weeks. Conventional therapy included: IV Dextran-40 (7 days), IV Ginkgo Biloba (14 days), oral Mecobalamin, and oral Yufeng Ningxin Dripping Pills.
  Arms: GAI Group
Drug: Conventional Therapy — Intravenous Dextran-40 (500 mL, daily for 7 days); Intravenous Ginkgo Biloba Extract (20 mL, daily for 14 days); Oral Mecobalamin tablets (0.5 mg, t.i.d.); Oral Yufeng Ningxin Dripping Pills (12 pills, t.i.d.) for 4 weeks. No sham injections were administered.
  Arms: Control Group

SUMMARY:
Sensorineural hearing loss (SNHL) accompanied by vertigo is a significant clinical challenge. Current conventional treatments often offer limited efficacy. This study evaluates the efficacy and safety of Gastrodin Acupoint Injection (GAI) as an adjunctive therapy based on the Traditional Chinese Medicine (TCM) theory of "treating both liver and heart." The trial compares the outcomes of patients receiving conventional therapy alone versus those receiving conventional therapy combined with GAI to determine improvements in auditory function, vestibular symptoms, and quality of life.

DETAILED DESCRIPTION:
SNHL with vertigo significantly impacts patients' quality of life, often leading to psychological distress. The pathophysiology involves vascular compromise and inner ear hypoxia. While conventional treatments (corticosteroids, vasodilators) are standard, their efficacy can be inconsistent. TCM suggests that disharmony in the Liver and Heart contributes to these symptoms. Gastrodin, extracted from *Gastrodia elata*, has neuroprotective and circulation-promoting properties. Acupoint injection combines pharmacology with meridian stimulation.

This prospective, randomized, controlled trial enrolled 100 eligible patients assigned to either a GAI group or a Control group. Both groups received a standard regimen (Dextran-40, Ginkgo Biloba Extract, Mecobalamin, and Yufeng Ningxin Dripping Pills). The GAI group additionally received gastrodin injections at specific acupoints: Local points (Tinggong, Tinghui, Yifeng) and Distal points (Baihui, Taichong, Neiguan, Shenmen) alternating every two days for 4 weeks. Efficacy is assessed via audiometry, dizziness scales, tinnitus questionnaires, psychological scales, and hemodynamic/biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Meeting diagnostic criteria for SNHL with vertigo.
* Disease course of 3 to 30 days.
* Pure Tone Average (PTA) at 0.5, 1, 2, and 4 kHz between 30 and 90 dB HL.
* Willingness to participate and sign informed consent.

Exclusion Criteria:

* Conductive or mixed hearing loss.
* Hearing loss due to trauma, tumor, or infection.
* Meniere's disease.
* Severe systemic diseases (cardiovascular, cerebrovascular, renal, or hepatic).
* Pregnancy or lactation.
* Known allergy to any of the study medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Pure Tone Average (PTA) | Baseline and Week 4
  Calculated as the average of air-conduction hearing thresholds at 0.5, 1, 2, and 4 kHz measured by audiometry.
Change in Dizziness Handicap Inventory (DHI) Score | Baseline and Week 4
  The DHI is a 25-item self-assessment questionnaire evaluating the functional, emotional, and physical impact of dizziness. The total score ranges from 0 to 100. Higher scores indicate greater perceived handicap and more severe dizziness symptoms.

SECONDARY OUTCOMES:
Change in Word Recognition Score (WRS) | Baseline and Week 4
  WRS assesses speech discrimination ability by measuring the percentage of words correctly identified from a phonetically balanced list at a comfortable listening level (40 dB above speech reception threshold). Scores range from 0% to 100%. Higher scores indicate better hearing function and speech understanding.
Change in Tinnitus Evaluation Questionnaire (TEQ) Score | Baseline and Week 4
  The TEQ is used to assess the severity and impact of tinnitus on daily life. The questionnaire consists of items related to tinnitus characteristics and patient distress. Higher total scores indicate more severe tinnitus symptoms and a greater negative impact on the patient.
Change in Hamilton Anxiety Scale (HAMA) Score | Baseline and Week 4
  The HAMA is a clinician-rated scale to measure the severity of anxiety symptoms. It consists of 14 items, each scored from 0 to 4. The total score ranges from 0 to 56, with higher scores indicating more severe anxiety.
Change in Hamilton Depression Scale (HAMD) Score | Baseline and Week 4
  The HAMD is a clinician-rated scale to measure the severity of depressive symptoms. It contains 17 or 24 items (depending on version used), with higher total scores indicating more severe depression.
Change in Mean Flow Velocity (Vm) of Middle Cerebral Artery | Baseline and Week 4
  Vm is measured using Transcranial Doppler (TCD) ultrasound in the middle cerebral artery. Measured in cm/s. In the context of ischemic pathology, an increase in Vm (within normal ranges) indicates improved cerebral blood perfusion.
Change in Pulsatility Index (PI) of Middle Cerebral Artery | Baseline and Week 4
  PI is a hemodynamic parameter measured using Transcranial Doppler (TCD) calculated as (Systolic Velocity - Diastolic Velocity) / Mean Velocity. It reflects downstream vascular resistance. A lower PI score indicates reduced vascular resistance and improved microcirculation.
Change in Serum Endothelin-1 (ET-1) Level | Baseline and Week 4
  Measurement of serum ET-1 levels via enzyme-linked immunosorbent assay (ELISA). ET-1 is a potent vasoconstrictor. Lower levels indicate reduced vasoconstriction and potentially improved microcirculation.
Change in Serum Nitric Oxide (NO) Level | Baseline and Week 4
  Measurement of serum NO levels via enzyme-linked immunosorbent assay (ELISA). NO is a vasodilator. Higher levels indicate improved vasodilation and endothelial function.
Incidence of Adverse Events | From enrollment through study completion, an average of 4 weeks
  Number of participants with adverse events including local pain, hematoma, or systemic reactions, assessed using CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhangjiakou, Zhangjiakou, Hebei, China